CLINICAL TRIAL: NCT06555250
Title: Interest of Bone Scintigraphy in the Search for Scaphotrapezoidal Osteoarthritis in the Context of Preoperative Assessment of Rhizarthrosi
Brief Title: Interest of Bone Scintigraphy in the Search for Scaphotrapezoidal Osteoarthritis
Acronym: PSR
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0207 - PSR
Record Dates: First submitted 2022-07-04; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Rhizarthrosis; Prosthesis Failure
Keywords: rhizarthrosis; bone scintigraphy
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rhizarthosis can be treated by prothesis of the carpo-metacarpal (CM) joint of the thumb. But, if the scaphotrapeziotrapezoid (STT) joint is also affected by arthrosis, treating the CM joint exclusively may result in partial pain relief. Thus, bone scintigraphy could identify early arthrosis of the STT joint when its appearance seems to be normal on planar radiography, suggesting another surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* failure of medical treatment of rhizarthrosis
* eligibility for prothesis
* no osteoarthritis of the STT joint on planar radiography
* no opposition from the patient

Exclusion Criteria:

* Refusal by a patient

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who beneficiate of a bone scintigraphy before arthroplasty for rhizarthrosis with failure medical treatment, without osteoarthritis of the STT joint on planar radiography
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Search for a statistically significant association between scintigraphic STT hyperfixation and residual pain after TM prosthesis for patients with no radiographically obvious STT involvement. | before surgery and 4 month after surgery
  STT scintigraphic hyperfixation and pain before surgery and 4 months after TM arthroplasty

SECONDARY OUTCOMES:
Search for an association between scintigraphic STT hyperfixation in quantitative analysis and residual pain after TM prosthesis for patients without advanced STT involvement on radiography. | before surgery
  SUVmax STT and pain before surgery and 4 months after TM arthroplasty
Assessing the involvement of other carpal joint compartments | before surgery
  Scintigraphic hyperfixation of other carpal joint compartments and pain before surgery and 4 months after TM arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement